CLINICAL TRIAL: NCT04330222
Title: Imaging the Arterial Pathology in Cerebral Small Vessel Disease Using 7 Tesla Magnetic Resonance Imaging
Brief Title: Cambridge 7 Tesla Cerebral Small Vessel Disease Study
Acronym: CamSVD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); Wolfson Brain Imaging Centre (Unknown)
Responsible Party: Principal Investigator, Christopher Osuafor, Study Co-ordinator and Co-investigator, University of Cambridge
Other Study IDs: A095132
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Cerebral Small Vessel Diseases; Cerebral Small Vessel Ischemic Disease; Lacunar Stroke
Keywords: Vascular Cognitive Impairment; Vascular Dementia; 7 Tesla Magnetic Resonance Imagine (7T MRI)
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Stroke, Lacunar; Dementia, Vascular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with lacunar stroke due to SVD
  Interventions: Diagnostic Test: 7 Tesla Magnetic Resonance Imaging; Other: Brief Memory and Executive Test
- Healthy stroke free volunteers
  Interventions: Diagnostic Test: 7 Tesla Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: 7 Tesla Magnetic Resonance Imaging — Diagnostic Imaging
Other: Brief Memory and Executive Test — Cognitive Assessment
  Groups: Patients with lacunar stroke due to SVD

SUMMARY:
CamSVD is jointly sponsored by the University of Cambridge and Cambridge University Hospitals NHS Foundation Trust.

We aim to explore and understand the underlying arterial pathology in Cerebral Small Vessel Disease (SVD) using ultra-high-field 7 Tesla MRI. We will optimise 7T Time-of-Flight MR angiography, blood suppressed MR sequence and phase-contrast (PC) MR angiography for visualization of perforating lenticulostriate arteries. This optimised sequences will be used to determine the range of arterial pathologies seen in individuals presenting with lacunar strokes. The pathologies of the perforating lenticulostriate arteries will be correlated with conventional clinical risk factors, cognition and radiological markers of SVD.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic lacunar stroke with corresponding lacunar infarct on MRI

Exclusion Criteria:

1. Unable/unwilling to consent;
2. Age<18;
3. Stroke aetiology due to cardio-embolism or large vessel disease;
4. Lacunar infarcts >1.5cm;
5. Severe stroke (NIHSS score ≥16);
6. Evidence of cortical infarct of any size;
7. Other major neurological diseases;
8. Severe systemic diseases such as heart failure, liver failure and kidney failure or any illness in the judgement of the investigator that could affect participation in the study;
9. MRI contraindications e.g. metal objects in or on the body, claustrophobia, pregnancy, known allergy to gadolinium containing contrast agent, impaired renal function with estimated glomerular filtration rate (eGFR) <59ml/min/1.73m2.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Lacunar Strokes due to Cerebral Small Vessel Disease
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2020-03-09 (Actual); Primary Completion 2024-01-12 (Estimated); Study Completion 2024-01-12 (Estimated)

PRIMARY OUTCOMES:
Range and pattern of pathology seen in the perforating arteries like presence or absence of focal atheroma and narrowing | March 2020-

SECONDARY OUTCOMES:
Differences in morphology of perforating arteries between SVD patients and healthy volunteers | March 2020-
Correlation of morphology of perforating arteries with cardiovascular risk factors and radiological markers of SVD | March 2020-

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Markus, FMedSci, Principal Investigator — University of Cambridge Department of Clinical Neurosciences
Locations (1):
- University of Cambridge, Cambridge, Cambridgeshire, United Kingdom